CLINICAL TRIAL: NCT06860516
Title: A Non-interventional Study of HLA-DRB1*04:01 Distribution in Adults With Recently Diagnosed Type 1 Diabetes (T1D)
Brief Title: HLA Demographics Study in Adults With Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: GentiBio, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: GNTI-T1D-HLA-1002
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type I
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a single blood draw for the analysis of HLA genotype of the study participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all participants: aged ≥ 18 to ≤ 45 years recently (within 2 months of the study visit) diagnosed with T1D
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — a blood draw for testing of HLA-DRB1*04:01

SUMMARY:
This is a study to evaluate the HLA-DRB1*04:01 genotype in adults that have been diagnosed with type 1 diabetes

DETAILED DESCRIPTION:
This is a non-interventional study to evaluate the distribution of human leukocyte antigen (HLA)-DRB1*04:01 genotype in participants that are recently (within 2 months of the study visit) diagnosed with T1D, with a single blood draw for the analysis of HLA genotype within the study participants. The study duration will be 24 hours and will include a single study visit for the collection of demographic data and a single blood draw, and a follow-up telephone call 24 hours after the study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged ≥ 18 to ≤ 45 years, with type 1 DM meeting American Diabetes Association criteria at diagnosis:

   1. Fasting glucose ≥ 126 mg/dL (7.0 mmol/L), or
   2. 2-hour oral glucose tolerance test plasma glucose ≥ 200 mg/dL (11.0 mmol/L), or
   3. Hemoglobin A1c ≥ 6.5%, or
   4. Random plasma glucose ≥ 200 mg/dL (11.1 mmol/L) (with documented classic hyperglycemia symptoms or hyperglycemic crisis).
2. Date of T1D diagnosis within 2 months of the study visit.
3. Able and willing to provide written, informed consent as approved by the institutional review board (IRB). Participants must be able to consent directly; no other person or guardian may consent for them in this study.

Exclusion Criteria:

1. Participant is an employee of, or an immediate family member of an employee, of the Sponsor, study site, or of a contractor/vendor who is involved in direct study conduct for this protocol.
2. Participant is unwilling or unable to comply with the study visit assessments.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will enroll up to 50 adults aged ≥ 18 to ≤ 45 years with recently (within 2 months of the study visit) diagnosed T1D who have met the American Diabetes Association T1D diagnosis criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
HLA DRB1*04:01 positive | Day 1
  to evaluate the frequency of adults with recently diagnosed type 1 diabetes that are HLA DRB1*04:01 positive at time of enrollment

SECONDARY OUTCOMES:
HLA-DRB1*04:01 genotype by ethnic and racial subgroups | Day 1
  to determine the distribution of HLA-DRB1*04:01 genotype in adults recently diagnosed with type 1 diabetes at the time of enrollment by ethnic and racial subgroups

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bach, MD, Study Director — GentiBio, Inc
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - University of Florida- Gainesville, Gainesville, Florida
  - Joslin Diabetes Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
will share study results through a publication or conference presentation
Supporting Information: CSR
Time Frame: within 6 months from study completion